CLINICAL TRIAL: NCT05993832
Title: Word Learning in Deaf Children Using Eye-tracking and Behavioral Measures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 4067E
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Deafness
Keywords: deafness; American Sign Language
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Referential cues to object (Experimental): Each object pair that is presented to the child is accompanied by 1) gaze only (3 trials); 2) novel label only (3 trials); or 3) conflicting gaze and novel label (3 trials)
  Interventions: Other: input cue

INTERVENTIONS:
Other: input cue — The object is labelled with 1) gaze only; 2) novel label only; or 3) conflicting gaze and novel label

SUMMARY:
Mutual exclusivity is a word learning constraint in which the learner assumes that a given word refers to only one category of objects. In spoken languages, mutual exclusivity has been demonstrated in monolingual children as young as 17 months and cross-linguistically, while multilingual learners show an attenuated mutual exclusivity bias. Mutual exclusivity has not been robustly demonstrated in deaf children acquiring American Sign Language (ASL). Further, it is unclear if mutual exclusivity applies to those learning both a signed and a spoken language. Like unimodal bilinguals, bimodal bilingual (BiBi) children learn two words for an object, but these words are separated by modality. A BiBi child could therefore assume that all objects have two words (like unimodal bilinguals) or that all objects have one spoken word and one sign (within-modality mutual exclusivity). The goals of the current study are to demonstrate mutual exclusivity in monolingual deaf children acquiring ASL, and to determine if BiBi deaf children utilize mutual exclusivity within each modality.

DETAILED DESCRIPTION:
The investigators will investigate how deaf children prioritize input cues to word meaning when linguistic cues (i.e. mutual exclusivity) and referential gaze are in conflict in a structured word learning task.

Participants: Deaf children (n=40) ages 24-60 months. Investigators will recruit 60 children to allow for 33% attrition. While the inclusion criteria are the same as other studies, here investigators do use spoken language exposure as a grouping variable, as follows: based on responses to the language background questionnaire regarding exposure to spoken English, participants will be grouped according to language use as monolingual ASL or bimodal bilingual (spoken English/ASL). Participants will be identified as bimodal bilingual is 1) the primary caregiver reports spoken English to communicate with their child (either alone or in conjunction with ASL), and 2) the primary caregiver reports that their child's ability to understand spoken English is at least a 3 on a Likert-type scale ranging from 0-5. Parents in this group will complete the short-form English CDI in addition to the ASL language measures.

Procedure: Participants will sit across a table from an experimenter who will present pairs of objects--one familiar, one novel--with one pair in each of nine trials (three per condition). The experimenter will prompt the participant to give them one of the toys, signing "I WANT YOU-GIVE-ME WHAT?" Then the experimenter will provide a cue; the child's selection will be recorded. In the gaze condition, the cue will be a gaze shift to the familiar object. In the mutual exclusivity condition, the cue will be a novel sign. In the conflict condition, both a gaze shift to the familiar object and a novel sign will be used. The trial order and object pair will be pseudo-randomly assigned.

Planned analysis: Investigators will use an omnibus mixed effects binomial model to determine how well condition and language environment predict the likelihood to select the novel object, with item and child as random factors.

ELIGIBILITY:
Inclusion Criteria:

* Deaf children ages 18-60 months
* born severely to profoundly deaf
* have either deaf or hearing parents
* communicate using American Sign Language
* have normal to corrected normal vision

Exclusion Criteria:

* Deaf children who have not been exposed to American Sign Language

Ages: 18 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Selected object | 10 seconds following experimenter prompt
  Children will select one of the two objects on the table in front of them. Their selection will be scored as correct or incorrect based on the target object.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Lieberman, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States